CLINICAL TRIAL: NCT03535974
Title: Evaluation of the Efficacy of a Supplement With Spirulina for Amelioration of Benign Thyroid Nodules
Brief Title: Efficacy of a Spirulina Supplement for Amelioration of Benign ThYroid Nodules
Acronym: ESSAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundatia Bio-Forum (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TiroNod
Record Dates: First submitted 2018-05-02; First posted 2018-05-24 (Actual); Results first posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Benign Thyroid Nodule

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preparation with Spirulina (Active Comparator): 6 weeks bid Preparation with Spirulina
  Interventions: Dietary Supplement: Preparation with Spirulina
- Placebo (Placebo Comparator): 6 weeks bid Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Preparation with Spirulina — Preparation with Spirulina to ameliorate the size of benign thyroid nodules
  Arms: Preparation with Spirulina
Dietary Supplement: Placebo — Placebo administration for 6 weeks bid
  Arms: Placebo

SUMMARY:
Clinical trial with a double-blind, placebo-controlled, crossover design; enrolls approximately 30 euthyroid patients with benign thyroid nodules, who will receive for 6 weeks a spirulina-based supplement, and for another 6 weeks placebo. Thyroid ecography will be performed three times for each patient, and blood tests including TSH, free T4, free T3 and ceruloplasmin/Copper will also be performed 3 times for each patient. It is expected that a decrease in the thyroid nodules occurs with the supplement administration. Compared with placebo there will be a decrease of at least 20% in the volume or the largest diameter of the nodules during the 6-week administration of the supplement.

DETAILED DESCRIPTION:
Clinical trial with double-blind, placebo-controlled, crossover design; enrolls approximately 30 euthyroid patients with benign thyroid nodules, who will receive for 6 weeks a spirulina-based supplement, and for another 6 weeks placebo.

* The sequence of administration supplement - placebo is unknown to the doctor or the patients
* The supplement and placebo are placed in identical capsules and vials by DVR Pharm
* The respective capsules are administered twice a day Thyroid ecography will be performed three times for each patient, and blood tests including TSH, free T4, free T3 and ceruloplasmin/Copper will also be performed 3 times for each patient.
* Echography and blood tests will be performed for each patient initially, after 6 weeks, and after 12 weeks It is expected that a decrease in the thyroid nodules occurs with the supplement administration.
* there will be a direct comparison of the nodules dimensions on the ecographic examinations, in millimeters, and of the blood levels of the molecules which reflect thyroid function

ELIGIBILITY:
Inclusion Criteria:

* euthyroid adults (normal TSH)
* no criteria for malignancy is present (size, fine needle aspiration, lymph nodules)
* no other medication/supplement administered for thyroid, no steroids, beta-blocker

Exclusion Criteria:

* suspicion of malignancy / shown
* autoimmune disease
* abnormal thyroid function
* Wilson disease
* contraception with intrauterine device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corin Badiu, M.D., Principal Investigator — Institutul Parhon
Locations (1):
- Fundatia Bio-Forum, Bucharest, București, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stancioiu F, Mihai D, Papadakis GZ, Tsatsakis A, Spandidos DA, Badiu C. Treatment for benign thyroid nodules with a combination of natural extracts. Mol Med Rep. 2019 Sep;20(3):2332-2338. doi: 10.3892/mmr.2019.10453. Epub 2019 Jul 1. PMID 31322200

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence AI-P: Active Ingredient (Spirulina) Then Placebo: Patients in this sequence first received 6 weeks the Active Ingredient (Spirulina) bid, and afterwards 6 weeks Placebo bid
- Sequence P-AI: Placebo Then Active Ingredient (Spirulina): Placebo administration for 6 weeks bid; afterwards Active Ingredient (Spirulina) for 6 weeks bid
- Sequence AI-AI (Active Ingredient, Then Active Ingredient): Patients receive Active Ingredient (AI) for 6 weeks bid, and afterwards Active Ingredient (AI) for 6 weeks bid
Period: First Intervention Weeks 0-6 (V1-V2)
Arm/Group | Sequence AI-P: Active Ingredient (Spirulina) Then Placebo | Sequence P-AI: Placebo Then Active Ingredient (Spirulina) | Sequence AI-AI (Active Ingredient, Then Active Ingredient)
Started | 14 | 19 | 5
Completed | 12 | 17 | 5
Not Completed | 2 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0
Period: Second Intervention Weeks 6-12 (V2-V3)
Arm/Group | Sequence AI-P: Active Ingredient (Spirulina) Then Placebo | Sequence P-AI: Placebo Then Active Ingredient (Spirulina) | Sequence AI-AI (Active Ingredient, Then Active Ingredient)
Started | 12 | 17 | 5
Completed | 12 | 17 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: For the primary outcome we compared the effect of the AI vs P after the initial 6 weeks of the study (V1-V2). For this we combined the AI-AI sequence and AI-P sequence in one arm, and compared with the P-AI sequence arm.
Groups:
- AI-P Sequence (12): Participants who received AI initially (first six weeks, V1 and V2) and P afterwards
- P-AI Sequence (17): Participants who received placebo (P) initially (first six weeks, V1 and V2) and AI afterwards
- AI-AI Sequence (5): Participants who received AI initially (first six weeks, V1 and V2) and AI afterwards
- Total: Total of all reporting groups
Arm/Group | AI-P Sequence (12) | P-AI Sequence (17) | AI-AI Sequence (5) | Total
Number analyzed (Participants) | 12 | 17 | 5 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 15 | 3 | 28
  >=65 years | 2 | 2 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.58 (7.03) | 52.12 (15.26) | 52.8 (15) | 53.44 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 16 | 3 | 29
  Male | 2 | 1 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 17 | 5 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Surface of Thyroid Nodules [Mean (Standard Deviation); unit: cm^2] — Surface of thyroid nodules in cm^2
  cm^2 | 4.18 (3.45) | 4.298 (3.01) | 5.18 (3.4) | 4.387 (3.139)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Area of Thyroid Nodules
Description: Size of the thyroid nodules is measured by ultrasound, two perpendicular diameters, same incidence and operator at V1 and V2 Area of nodules is calculated as the product of the two diameters
Time Frame: after 6 weeks of administration of the supplement and placebo
Population: Effects of AI vs P between the two arms is calculated after the first 6 weeks (V1-V2, AI vs P). After 12 weeks (V1-V3) patients in each arm/sequence receive the same treatment in a different sequence (AI+P; vs P+AI) and no difference is expected.
  A second outcome compares results of all administrations of 6 weeks each of AI (39) and P (29)
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Preparation With Spirulina: 6 weeks bid Preparation with Spirulina
  Preparation with Spirulina: Preparation with Spirulina to ameliorate the size of benign thyroid nodules decrease of 19.88% (mean) +/- 15.55 (SD)
- Placebo: 6 weeks bid Placebo
  Placebo: Placebo administration for 6 weeks bid decrease of 9.21% (mean) +/- 14.29 (SD)
Arm/Group | Preparation With Spirulina | Placebo
Number analyzed (Participants) | 17 | 17
percentage change | -19.98 (15.55) | -9.31 (14.29)
Statistical Analysis 1: Comparison: Preparation With Spirulina vs Placebo; Test type: Other; p = 0.047, t-test, 2 sided; Mean Difference (Final Values) = 10.57, Standard Error of Mean 5.122

2. Post Hoc Outcome: Mean Change in Nodule Areas, All Administrations of 6 Weeks Each (n=68), AI (n=39) Versus P (n=29)
Description: Mean modification in the area of the nodules in cm^2, calculated as the difference between the initial and final nodule area after 6 weeks of administration of either AI (total 39 administrations) or P (total 29 administrations), and standard deviation
Time Frame: after 12 weeks of administration of the supplement and placebo
Population: The total number (instances) of 6 weeks administrations of either AI (n=39) or P (n=29)
Measure: Mean (Standard Deviation); unit: cm^2
Groups:
- All AI Administrations (n=39): Number of all 6 weeks administrations of AI in all 34 patients and all sequences (AI-P, AI-AI, and P-AI)
- All P Administrations (n=29): Number of all 6 weeks administrations of P in all 34 patients and all sequences (AI-P and P-AI)
Arm/Group | All AI Administrations (n=39) | All P Administrations (n=29)
Number analyzed (Participants) | 39 | 29
cm^2 | 0.611 (0.933) | 0.178 (0.515)

ADVERSE EVENTS:
Time Frame: 6 months
Description: One patient who was on multiple medications at enrollment developed a generalized skin eruption with moderate prurit after a few days with the study substance; she interrupted the administration after talking with the investigator and afterwards it was revealed that she was taking placebo All participants who completed the study (n=34) received the AI (active ingredient) and 5 patients out of the 34 (n=29) received the AI-AI sequence, so that only 29 patients received placebo (P)
Groups:
- Preparation With Spirulina: 6 weeks bid Preparation with Spirulina
  Preparation with Spirulina: Preparation with Spirulina to ameliorate the size of benign thyroid nodules
  0 adverse reactions
- Placebo: 6 weeks bid Placebo
  Placebo: Placebo administration for 6 weeks bid
  One patient had a severe allergic reaction while she was on placebo and multiple other medications and withdrew from the study
Arm/Group | Preparation With Spirulina | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/34 | 1/29
Other Adverse Events (participants affected / at risk) | 0/34 | 1/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preparation With Spirulina (N=34) | Placebo (N=29)
allergic reaction while on placebo (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preparation With Spirulina (N=34) | Placebo (N=29)
allergic reaction while on placebo (Immune system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT03535974/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT03535974/ICF_001.pdf